CLINICAL TRIAL: NCT05256758
Title: The Effect of Altering Myocardial Lipid Content on Cardiac Physiology in Patients With Aortic Stenosis
Brief Title: Oxford - Fibrates in Aortic Stenosis
Acronym: OxFAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OxFAST
Record Dates: First submitted 2022-01-20; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Fenofibrate; Placental Lactogen

STUDY DESIGN:
Intervention Model Description: Randomised double-blind placebo controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomised double-blind placebo controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OxFAST Fibrate group (Experimental): 49 patients randomised to receive fenofibrate 200mg capsules.
  Interventions: Drug: Fenofibrate Capsules
- OxFAST placebo group (Placebo Comparator): 13 patients randomised to receive placebo will act as controls.
  Interventions: Drug: Placental Lactogen

INTERVENTIONS:
Drug: Fenofibrate Capsules — 49 patients randomised to receive fenofibrate for 6 months.
  Other Names: Fenofibrate
  Arms: OxFAST Fibrate group
Drug: Placental Lactogen — 13 patients randomised to receive placebo for 6 months.
  Arms: OxFAST placebo group

SUMMARY:
Aortic stenosis (AS) is characterised by left ventricular (LV) hypertrophy and altered myocardial substrate metabolism. Peroxisome proliferator-activated receptor (PPARα), a regulator of lipid metabolism is deactivated in pressure overload hypertrophy such as in AS and can lead to dysregulation of fatty acid oxidation, myocardial triglyceride accumulation (steatosis) and lipotoxicity. The investigators propose a proof-of-concept study to investigate the effect of altering myocardial triglyceride (MTG) using a PPARα agonist, fenofibrate on cardiac physiology in patients with asymptomatic moderate-severe AS. The primary endpoint is a change in MTG assessed by magnetic resonance spectroscopy at baseline and after 6 months of treatment. Exploratory endpoints are changes in cardiac physiology including myocardial deformation (strain) as assessed by cardiac magnetic resonance imaging. The investigators hypothesise that pharmacological reduction of MTG with a PPARα agonist will result in steatosis regression and changes in cardiac physiology.

DETAILED DESCRIPTION:
This is a single-centre, proof-of-concept study to investigate the effect of altering MTG content using fenofibrate on cardiac physiology in patients with asymptomatic moderate-severe AS. All patients will participate in a randomised, double-blind, placebo- controlled design for 6 months. AS will be graded according to the British Society of Echocardiography's transthoracic echocardiography guidelines. Sixty two eligible patients will be recruited in total, of which forty nine patients will be randomised to receive 200 mg daily oral fenofibrate and thirteen patients will receive matching placebo for 6 months. All patients will undergo 1H-MRS to assess MTG, 31P-MRS to assess myocardial energetic (Phosphocreatine-to-ATP ratio - PCr/ATP), standard cardiac magnetic resonance imaging to assess LV strain, LV mass, late gadolinium enhancement (fibrosis), physiological exercise assessments to measure maximum oxygen consumption (VO2 max) and 6-minute walking distance. Bloods will be drawn for cholesterol, renal and liver function, glucose and free fatty acids. All tests will be done at baseline and after 6 months' treatment with fenofibrate/placebo.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic moderate to severe AS (with at least two of the following: aortic valve area <1.5 cm2, peak pressure gradient >36 mmHg or mean pressure gradient >25 mmHg)
* Not planned aortic valve replacement or transcatheter aortic valve implantation (TAVI)
* Age >18
* No other significant valvular pathology
* No contraindication to magnetic resonance imaging.

Exclusion Criteria:

* Known coronary artery disease, history of angina, myocardial infarction or presence of regional wall motion abnormalities
* Other underlying cardiomyopathy
* Left ventricular ejection fraction<50%
* Uncontrolled hypertension
* Diabetes Mellitus
* Liver impairment
* Pregnancy and lactation
* Body mass index >35 kg/m2
* Renal impairment (eGFR<30 ml/min)
* Intolerance to or concurrent use of fibrates or PPARα agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial triglyceride (MTG) content as assessed by cardiac magnetic resonance (CMR) spectroscopy | 6 months
  All participants will undergo blood tests (full blood count, renal and liver function, lipid profile, free fatty acids and NT- proBNP), CMR cine imaging for assessment of cardiac volumes, function including strain (myocardial tagging), aortic valve imaging and late gadolinium enhancement will be undertaken.
  MTG will be assessed using cardiac 1H-MRS (proton spectroscopy), which utilises the abundant hydrogen (1H) protons. For 1H-MRS, data are typically acquired at breath hold during diastole from a single voxel (14-16mL) localised in the myocardial septum and take 10-15 minutes to acquire. Myocardial lipid content is calculated as myocardial lipid/water ratio and expressed as percentage.
  It is hypothesised that Fenofibrate, PPAR alpha agonist will shift the cardiac metabolism back to mainly using free fatty acids and hence the investigators may see a reduction in myocardial lipid content.

SECONDARY OUTCOMES:
Change in myocardial energetics (PCr/ATP ratio) as assessed by Phosphorous magnetic resonance spectroscopy | 6 months
  31P-MRS (Phosphorous Spectroscopy) allows the in vivo quantification of phosphorus (31P)-containing metabolites involved in energy metabolism, such as Phosphocreatine and ATP (Adenosine Triphosphate). PCr/ATP ratio is a reliable indicator of myocardial energetics. It is hypothesised that fenofibrate will increase fatty acid metabolism in the heart and subsequently improve the energetic status of the heart.
Change in left ventricular function measured using CMR imaging | 6 months
  The investigators will assess the effect of altering cardiac metabolism using Fenofibrate and study its effect on cardiac physiology, mainly left ventricular function using CMR imaging. Strain assessment using myocardial tagging analysis will be used to detect subclinical dysfunction. The strain values are expressed as percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmod, Principal Investigator — University of Oxford
Locations (1):
- OUH NHS trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT05256758/Prot_SAP_000.pdf